CLINICAL TRIAL: NCT03538366
Title: Fecal Microbiota Transplantation for the Treatment of Chronic Pouchitis
Brief Title: Fecal Microbiota Transplantation for Chronic Pouchitis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aalborg University Hospital (Other)
Responsible Party: Principal Investigator, Ole Thorlacius-Ussing, MD, DMSc, Professor of Surgery, MD, DMSc, Professor of Surgery, Aalborg University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FMT and Pouchitis
Record Dates: First submitted 2018-05-11; First posted 2018-05-29 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Ulcerative Colitis; Pouchitis
Keywords: Ulcerative Colitis; Inflammatory bowel disease; Pouchitis; Fecal microbiota transplant; Fecal microbiota treatment
MeSH Terms: conditions — Colitis, Ulcerative; Pouchitis; Inflammatory Bowel Diseases

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Donor FMT (Experimental): Fecal transplant from unrelated, healthy volunteers
  Interventions: Other: Donor FMT

INTERVENTIONS:
Other: Donor FMT — Fecal transplant from unrelated, healthy donors using enemas

SUMMARY:
Patients with chronic pouchitis are treated with fecal transplant from several unrelated, healthy donors. The treatment consists of enemas of 100 mL fecal suspension, applied for 14 consecutive days.

DETAILED DESCRIPTION:
Background:

The surgical treatment of choice for the treatment of medically refractory ulcerative colitis (UC) is restorative ileal pouch-anal anastomosis (IPAA), in which the patient retains fecal continence following colonectomy, by subsequent anastomosis of the terminal ileum and the rectum.

Up to 25% of patients with UC will undergo IPAA surgery. The most common complication following the procedure is inflammation of the pouch (pouchitis), which is seen in up to 50% of patients within the first five years of surgery. Of these patients, 10-20% will develop a chronic inflammatory condition. The clinical symptoms of pouchitis include diarrhea, rectal bleeding, stomach cramps, general malaise and reduced quality of life. Endoscopic findings include mucosal edema, granulations, and ulcerations with mucosal frailty. In most cases, a causative microorganism is not identified, although infection with Clostridium difficile or Cytomegalovirus (CMV) have been reported.

The most common treatment of pouchitis is empiric antibiotics, usually quinolones and metronidazole, or a combination of both. Following complications, removal of the pouch can become a last resort, and chronic pouchitis is the leading indication for 10% of these operations.

The composition of microbes in the gut is known to be a key factor in the homeostasis of the intestine, and plays a central role in the development of CIBD. Different single microorganisms have previously been suggested as playing an important role in this development, including: Mycobacterium avium, Escherichia coli and Clostridium difficile, that all have invasive capabilities. Several studies have investigated the connection between the composition of microbes in the gut and development of pouchitis finding an increasing evidence for a link between dysbiosis and pouchitis.

Method:

Patients with chronic pouchitis are treated with fecal transplants from unrelated, healthy donors. The fecal transplant is from several healthy donors. The treatments are applied as enemas of 100 ml suspension for 14 consecutive days.

Prior to treatment, pouchitis activity is graded using the pouchitis disease activity index (PDAI) based on symptoms, endoscopic and histological criteria. Patients will also complete self-reported questionnaires regarding pouch function, quality of life and sexuality.

Patients are evaluated using the PDAI score 30 days following treatment together with the self-reported questionnaires. Longterm follow up is evaluated up to 6 months following FMT.

Screening of FMT donors:

1. Questionaire regarding possible contagious infectious diseases, followed by interview with principal investigator.
2. Blood test for: inflammatory parameters: CRP, leucocyte count, HIV 1+2 antigen, Hepatitis A, B and C, CMV, EBV and HbA1c
3. Fecal samples:

   1. Calprotectin
   2. Pathogenic bacteria (Salmonella, Campylobacter, Yersinia, Shigella), Vibrio, toxin-producing E. coli.
   3. Parasites, giardia spp. and cryptosporidium spp.
   4. Adenovirus, enterovirus, parechovirus
   5. Clostridium difficile
   6. Vancomycin-resistent Enterococcus faecalis and Enterococcus faecium, carbapenemase-producing enterobacteria and ESBL-producing E.coli.

FMT donor exclusion criteria are:

* Age <20 or >65
* BMI <18.5 or > 28.0 kg/m2
* Known chronic inflammatory bowel disease, celiac disease, rheumatoid arthritis or other autoimmune disease, sclerosis, psoriasis, previous extensive bowel surgery
* In the previous 6 months:
* Diarrhea > 3 days in one week or bloody stools
* Treatment with antibiotics
* Risk of sexually transmitted disease, tattoos, piercings, travel to areas with high endemic transmission of infectious diseases or resistants microbes.

ELIGIBILITY:
Inclusion Criteria:

* minimum 18 years old, pouch > 1 year
* at least three pouchitis events in the past year
* antibiotic treatment for pouchitis at least one time in the past year

Exclusion Criteria:

* immunosuppression, pregnancy, detection of specific pathogens in stool

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2018-05-15 (Actual); Primary Completion 2019-05-01 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Cure 30 days following FMT treatment | 30 days
  PDAI < 7

SECONDARY OUTCOMES:
Changes of the microbiota | 30 days
  Changes in diversity of gut microbiota after FMT assessed by Shannon index
Clinical response 30 days after FMT treatment | 30 days
  Decrease from baseline PDAI > 2 points
Histological remission following PDAI | 30 days
  Remission of microscopic inflammation
Improvement of pouch function | 30 days
  Improvement of the self-reported questionnaire
Improvement of quality of life | 30 days
  Improvement of the self-reported questionnaire
Improvement of sexuality | 30 days
  Improvement of the self-reported questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Ole Thorlacius-Ussing, Professor, Study Director — Aalborg University Hospital, Aalborg University
Locations (1):
- Research Unit, Department of Gastrointestinal Surgery, Aalborg, Denmark

REFERENCES:
- [Background] Becker JM. Surgical therapy for ulcerative colitis and Crohn's disease. Gastroenterol Clin North Am. 1999 Jun;28(2):371-90, viii-ix. doi: 10.1016/s0889-8553(05)70061-3. PMID 10372273
- [Background] Onaitis MW, Mantyh C. Ileal pouch-anal anastomosis for ulcerative colitis and familial adenomatous polyposis: historical development and current status. Ann Surg. 2003 Dec;238(6 Suppl):S42-8. doi: 10.1097/01.sla.0000098115.90865.16. PMID 14703744
- [Background] Lovegrove RE, Tilney HS, Heriot AG, von Roon AC, Athanasiou T, Church J, Fazio VW, Tekkis PP. A comparison of adverse events and functional outcomes after restorative proctocolectomy for familial adenomatous polyposis and ulcerative colitis. Dis Colon Rectum. 2006 Sep;49(9):1293-306. doi: 10.1007/s10350-006-0608-0. PMID 16830218
- [Background] Sandborn WJ. Pouchitis following ileal pouch-anal anastomosis: definition, pathogenesis, and treatment. Gastroenterology. 1994 Dec;107(6):1856-60. doi: 10.1016/0016-5085(94)90832-x. No abstract available. PMID 7958702
- [Background] Shen B. Diagnosis and treatment of patients with pouchitis. Drugs. 2003;63(5):453-61. doi: 10.2165/00003495-200363050-00002. PMID 12600225
- [Background] Shen B, Achkar JP, Lashner BA, Ormsby AH, Remzi FH, Brzezinski A, Bevins CL, Bambrick ML, Seidner DL, Fazio VW. A randomized clinical trial of ciprofloxacin and metronidazole to treat acute pouchitis. Inflamm Bowel Dis. 2001 Nov;7(4):301-5. doi: 10.1097/00054725-200111000-00004. PMID 11720319
- [Background] Sandborn WJ, Pardi DS. Clinical management of pouchitis. Gastroenterology. 2004 Dec;127(6):1809-14. doi: 10.1053/j.gastro.2004.10.011. No abstract available. PMID 15578518
- [Background] Khan KJ, Ullman TA, Ford AC, Abreu MT, Abadir A, Marshall JK, Talley NJ, Moayyedi P. Antibiotic therapy in inflammatory bowel disease: a systematic review and meta-analysis. Am J Gastroenterol. 2011 Apr;106(4):661-73. doi: 10.1038/ajg.2011.72. Epub 2011 Mar 15. PMID 21407187
- [Background] Tulchinsky H, Hawley PR, Nicholls J. Long-term failure after restorative proctocolectomy for ulcerative colitis. Ann Surg. 2003 Aug;238(2):229-34. doi: 10.1097/01.sla.0000082121.84763.4c. PMID 12894016
- [Background] Angriman I, Scarpa M, Castagliuolo I. Relationship between pouch microbiota and pouchitis following restorative proctocolectomy for ulcerative colitis. World J Gastroenterol. 2014 Aug 7;20(29):9665-74. doi: 10.3748/wjg.v20.i29.9665. PMID 25110406